CLINICAL TRIAL: NCT03260556
Title: Pirfenidone for Progressive Fibrotic Sarcoidosis
Acronym: PirFS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Robert P Baughman, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-5706
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Sarcoidosis, Pulmonary
Keywords: pulmonary fibrosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pirfenidone (Active Comparator): Pirfenidone titrated to three 267 mg tablets three times a day
  Interventions: Drug: Pirfenidone
- Placebos (Placebo Comparator): Placebo titrated to three tablets three times a day
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Pirfenidone — Increasing doses
  Other Names: esbriet
  Arms: Pirfenidone
Drug: Placebos — Increasing doses
  Other Names: placebo
  Arms: Placebos

SUMMARY:
Study comparing pirfenidone versus placebo for patients with advanced fibrotic sarcoidosis

DETAILED DESCRIPTION:
Patients who meet the inclusion and exclusion criteria will be randomized to be treated with either placebo or pirfenidone at the current approved dosage for idiopathic pulmonary fibrosis at a 2:1 pirfenidone to placebo ratio. Patients treated with pirfenidone will be titrated using the following schedule:

One 267 mg capsules three times a day for two weeks. Two 267 mg capsules three times a day for two weeks Three 267 mg capsules three times a day thereafter Patients will be instructed to take all doses of medication with food. Dosage will be titrated on an individual basis depending on patient tolerance of medication.

Those randomized to placebo will receive the same schedule using placebo tablets.

Block randomization will be done at each site. Liver function tests will be evaluated as listed above. If the patient has an abnormal liver function test, then the dose will be adjusted per the company's protocol for commercial drug.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoidosis
* Pulmonary function testing with a Composite Physiologic Index (CPI) score of greater than 40
* Patient must have evidence of >20% fibrosis on high resolution cat scan
* Patients must be on a stable prednisone therapy for sarcoidosis for at least two months and no change in other immunosuppressives in the two months prior to entry into study
* Age greater than 18 and less than 90.
* Able to provide written informed consent for participation in the study

Exclusion Criteria:

* Patients receiving therapy for precapillary pulmonary hypertension.
* Patients with liver disease Childs class 3 or 4
* Patients with a left ventricular ejection fraction of less than 40%
* Patients receiving more than 20 mg prednisone daily or its equivalent
* Patients with massive hemoptysis within prior three months. Patients with mycetomas are eligible as long as no massive hemoptysis in prior three months.
* Patients with clinically important co-existing disease which in the opinion of the investigator is likely to affect patient's chance for survival during the course of the study
* Patient who is pregnant, lactating, intending to become pregnant during the study, or child bearing capacity who is not willing to use appropriate birth control methods approved by investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Time until clinical worsening (TCW) | two years
  TCW

SECONDARY OUTCOMES:
Change in forced vital capacity (FVC) | two years
  Change in forced vital capacity
Change in CPI | two years
  Change in composite physiologic index

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
no plans yet